## **STUDY INFORMATION SHEET**

Version 3. Date: 29/05/2025

Principal Investigator: Alba Sierra Yagüe

Es tu juego: Decide Bien [It's Your Game: Keep It Real]. Cultural Adaptation, Validation, and Evaluation of the Programme for Promotion of Healthy AffectiveSexual Behaviours in Adolescents

This document is to inform you about a study being carried out by a research group from the University of Granada and the University of Seville, in which your son/daughter is invited to participate. The study has been approved by the Provincial Research Ethics Committee of Granada under code 202499906944441.

The sole purpose is to ensure that you receive accurate and sufficient information to assess and decide whether you wish to give your consent for your child's participation in this study. Please read this information sheet carefully and feel free to ask any questions you may have.

## STUDY OBJECTIVE

The objective of the study is to carry out the cultural adaptation of the program *It's Your Game: Keep it Real (IYG)*, which aims to prevent risky sexual and affective behaviors in adolescents. The IYG program consists of 12 lessons, each lasting 45 minutes. These lessons are designed to help adolescents identify their personal norms and boundaries regarding sexuality, recognize situations that might challenge those boundaries, and develop refusal skills to maintain them. The program also addresses other topics of interest such as characteristics of healthy and unhealthy relationships, friendships, anatomy and reproduction, the social, emotional, and physical consequences of sexual activity, the consequences of teenage pregnancy and sexually transmitted infections (STIs), condom and contraceptive use, and communication skills.

This adaptation will involve your child completing the 12 lessons (two per week over six weeks) that make up the IYG program, as well as completing a series of questionnaires to assess the usability of the program in Spain (including ease of use, comprehension, acceptability, aspects most liked, and suggestions for improvement).

Participation is entirely **VOLUNTARY AND ANONYMOUS**, and you may withdraw your consent at any time, without providing any explanation and without this affecting the care your child will receive.

In all cases, **CONFIDENTIALITY** of the collected data will be maintained in accordance with the European Union General Data Protection Regulation (GDPR) 2016/679 and the Spanish Organic Law on the Protection of Personal Data and Guarantee of Digital Rights (LOPD-GDD) 3/2018, of December 5.

The results of the study may be shared with the scientific community through presentations, conferences, and/or publications.

Thank you in advance for your collaboration in this study.

For any **ADDITIONAL INFORMATION**, please contact the principal investigator of this study, Alba Sierra Yagüe (asierra.mn.ics@gencat.cat).

## **INFORMED CONSENT FORM**

| <b>Project Title:</b> "Es tu juego: Decide Bien [It's Your Game: Keep It Real]. Cultural Adaptation, Validation, and Evaluation of the Programme for Promotion of Healthy Affective-Sexual Behaviours in Adolescents" |
|---|
| Participant's Full Name: Legal Representative's Full Name: ID Number (DNI/NIE): |
| CONSENT: I,, declare under my responsibility that I have read and understood the Information Sheet, of which I have been given a copy. |
| I have received sufficient information about my child's participation in the project and about the use of his/her personal data and associated information. I have been able to ask questions about the information provided and to speak with the principal investigator, who has answered all the questions I have asked. |
| <ul> <li>I understand that my child's participation is voluntary.</li> </ul> |
| <ul> <li>I understand that all my child's data will be treated confidentially.</li> </ul> |
| I understand that participation can be withdrawn: |
| o At any time. |
| <ul> <li>Without having to provide any explanation.</li> </ul> |
| Therefore, having read the information and conditions of the study: Yes, I freely give my consent for my child to participate in the study. No, I do not give my consent. In, on the day of 202 |
| Signature of legal guardian |
| WITHDRAWAL OF INFORMED CONSENT |
| If you decide to withdraw participation from the study, please complete the following information and send it by email to: <a href="mailto:asierra.mn.ics@gencat.cat">asierra.mn.ics@gencat.cat</a> |
| I, parent/guardian of the minor with ID (DNI/NIE – last 4 digits and letter) (e.g., 2795D), hereby declare that: |

| I revoke the informed | l consent prev | iously granted, | and from this mor | nent, I withdraw |
|---|---|---|---|---|
| permission for the use of my child's data in this research. | | | | |
| In | _, on the | _ day of | 202 | |